CLINICAL TRIAL: NCT06521229
Title: An Ambispective Observational Multicenter Registry of Patients With Uncontrolled Asthma in the Population of the Russian Federation
Brief Title: Clinical& Demographic Profiles of patIents With unControllEd Asthma in Russia: Multi-center oBsErvational ReGistry Study
Acronym: ICEBERG
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00206
Record Dates: First submitted 2024-06-21; First posted 2024-07-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Uncontrolled Asthma
Keywords: uncontrolled asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-centre, non-interventional, observational, ambispective registry. Planned study population consists of 9 000 adult patients with uncontrolled asthma receiving treatment according to standard of care (except biologics). Planned number of study site is 70 outpatient centers with experience of uncontrolled asthma treatment in about 50 regions of Russia (in order to describe characteristics of patients with uncontrolled asthma in different regions in the most comprehensive way).

DETAILED DESCRIPTION:
There are limited epidemiological data of the patients with uncontrolled asthma in Russia. The systematic information about complications and comorbidities, about the treatment approaches and their effectiveness in the Russian population is also absent.

The observational registry is really important to describe the epidemiological characteristics of the disease and to analyse the clinical characteristics of the various subgroups of patients. This is an excellent starting point to be able to investigate the characteristics of the disease in detail.

The Russian Federation consists of 85 regions with a total population of more than 145 million people. The regions differ in ethnic composition, age, gender, climate, ecology, economic level, prevalence of asthma in general and uncontrolled asthma in particular.

Thus, there is a need to perform a large-scale observational registry in regions of the country with a sufficient size of population to obtain information on uncontrolled asthma epidemiology, clinical and demographic characteristics, to describe main clinical outcomes and evaluate existing associations between observed treatment patterns and clinical outcomes in real clinical practice in patients with uncontrolled asthma not receiving biologic therapy.

Trial will have ambispective design and will include 2 visits for obtaining the patient's demographic and clinical data. To allow wide data coverage the study will involve at least 50 regions of Russian Federation; in each region 200 patients will be recruited. The total size of study population will be 9 000 patients.

All data will be collected during 2-3 visits carried out according to routine clinical practice for observation and treatment of patients with uncontrolled asthma. At visit 1, baseline data of 52 weeks prior to inclusion will be collected by physician based on the patient's medical records and interview during the visit. Visit 2 (final visit) will be conducted after 12 weeks (±7 days) in order to collect follow-up data which coincides with the recommended dates. Information on changes in the treatment of uncontrolled asthma and on clinical outcomes will be collected.

For the cohort of patients receiving fixed-dose combination budesonide/salbutamol on Visit 2, an additional follow-up visit (Visit 3) will be conducted in 12 weeks (±14 days) after Visit 2, in order to collect data which coincides with the recommended dates. Information on changes in the treatment of uncontrolled asthma and on clinical outcomes will be collected. It is planned to enroll 500 patients receiving fixed-dose combination budesonide/salbutamol on Visit 2, to whom the follow-up visit (Visit 3) will be conducted.

This non-interventional study does not imply any intervention into a routine clinical practice, and does not provide for any diagnostic and therapeutic procedures other than those used in routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of inclusion;
2. Signed and dated written informed consent in accordance with ICH GCP and local law prior to inclusion in the study;
3. Patients with diagnosis of uncontrolled mild and moderate asthma (according to Global Initiative for Asthma (GINA) score);
4. Patients with the availability of at least 52 weeks of follow-up data (prior to inclusion) in the medical records.

Exclusion Criteria:

1. Patients with severe asthma or/and patients receiving any biological therapy currently or within 52 weeks prior to inclusion;
2. Presence of chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (ILF) currently or in the anamnesis;
3. The participation in any clinical study currently or within 52 weeks prior to inclusion;
4. An acute or chronic disease that, as deemed by Investigator, limits the ability of patients to participate in this study or could influence the interpretation of the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 10 000 adult patients with confirmed diagnosis of uncontrolled mild and moderate asthma who receive medical treatment (excluding biological therapy) and are monitored and treated by pulmonologists or allergologists in approximately 70 clinical centers in about 50 regions of Russia
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
To describe the baseline demographic characteristics of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 12 weeks (also 52 weeks of retrospective data before visit 1)
  1. Mean age at the inclusion into the study;
  2. Mean age at the primary asthma diagnosis;
  3. Proportion of men and women;
  4. Mean body mass index (BMI);
  5. Proportion of patients with overweight (BMI ≥25 kg/m2);
  6. Proportion of patients with each educational status (higher, secondary special, secondary general);
  7. Proportion of patients from each residential region of Russia;
  8. Proportion of patients with negative lifestyle factors:
     1. Proportion of patients with history of smoking/current smokers - applicable to smoking tobacco and electronic cigarettes (vapes);
     2. Mean smoking index (pack-years) for current (tobacco) smokers;
     3. Mean duration of smoking (years) for current e-cigarette (vape) smokers;
     4. Proportion of patients with a history of alcohol abuse/current alcohol abuse;
     5. Proportion of patient with limitation of physical activity.
  9. Proportion of patients with chronic rhinosinusitis with nasal polyps;
  10. Proportion of patients with different comorbidities
To describe the baseline clinical characteristics of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  16. Mean FeNO (parts per billion (ppb)) (in case of availability of laboratory data)
To characterise the profile of routine therapy used for outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks (also 52 weeks of retrospective data before visit 1)
  17. Proportion of patients receiving different classes of drugs for treatment of asthma as reliever and maintenance therapy:
  1. SABA alone;
  2. ICS alone;
  3. LABA alone;
  4. ICS and LABA;
  5. ICS and SABA;
  6. ICS and LABA plus:
  a) SABA; b) LAMA; c) LTRA; d) Theophylline; e) Macrolide antibiotics. f) ICS and LABA (MART therapy) 18. Proportion of patients with ICS-containing therapy as reliever and as maintenance at baseline; 19. Proportion of patients using SABA reliever for symptoms more than two times a week at baseline; 20. Proportion of patients receiving OCS: intermittent (for exacerbations) / regularly (in the frame of basic therapy); 21. Mean number of OCS treatment courses; 22. Median daily dose in case of regular OCS use; 23. Median cumulative OCS exposure for exacerbations 24. Median cumulative OCS exposure in the frame of basic therapy; 25. Mean baseline parameters of lung function (in case of availability of spirometry data)
To describe the baseline eosinophils blood count of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  12. Proportion of patients with different levels of eosinophils blood count (in case of availability of laboratory data):
  1. <150 cells/μl;
  2. ≥150 cells/μl;
  3. ≥300 cells/μl.
To describe the baseline mean eosinophils count in sputum of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  13. Mean eosinophils count in sputum (cells per high power field) (in case of availability of laboratory data);
To describe the baseline mean total IgE of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  14. Mean total IgE (IU/ml) (in case of availability of laboratory data);
To describe the baseline Proportion of patients with different levels of total IgE of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  15. Proportion of patients with different levels of total IgE (in case of availability of laboratory data)
To describe the baseline Mean eosinophils blood count of outpatients with uncontrolled asthma in the Russian Federation in all patients and in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 12 weeks and 52 weeks of retrospective data before visit 1
  11. Mean eosinophils blood count (cells/μl) (in case of availability of laboratory data);

SECONDARY OUTCOMES:
1. Proportion of patients with controlled and partly controlled asthma at visit 2 in all patients and in the cohort of patients receiving FDC budesonide/salbutamol | 12 weeks (also 52 weeks of retrospective data before visit 1)
  according to GINA (Global Initiative for Asthma) score. GINA assessment of asthma control consists of 4 questions, the higher the score the worse asthma control is.
2. Proportion of patients with changes of inhaled asthma therapy occurred from baseline to visit 2 (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | 12 weeks (also 52 weeks of retrospective data before visit 1)
  1. Change of reliever;
  2. Change of dose of reliever;
  3. Change of number of reliever inhalations per day;
  4. Change of basic therapy drug;
  5. Change of dose of basic therapy drug;
  6. Change of number of basic therapy drug inhalations per day;
  7. Change of ICS;
  8. Dose of ICS increased;
  9. Changes of another drug for maintenance therapy.
  10. Change in the type of drug delivery within the same INN (e.g. from capsule to powder or from aerosol to powder, etc.)
3. Proportion of patients with OCS prescription occurred from baseline to visit 2 (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | 12 weeks (also 52 weeks of retrospective data before visit 1)
  for patients already used OCS at baseline dose change will be evaluated
4. Proportion of patients with ICS-containing therapy as reliever and as maintenance at visit 2 | 12 weeks (also 52 weeks of retrospective data before visit 1)
  (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol)
5. Proportion of patients using SABA reliever for symptoms more than two times a week at visit 2 (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | 12 weeks (also 52 weeks of retrospective data before visit 1)
  1. Proportion of patients using SABA reliever for symptoms more than two times a week at visit 1;
  2. Proportion of patients using SABA reliever for symptoms more than two times a week at visit 2;
  3. Proportion of patients who were not receiving SABA for symptom relief more than two times a week at baseline at Visit 1 and who began receiving SABA for symptom relief more than two times a week at Visit 2
6. Proportion of patients experiencing 0, 1, 2, ≥3 severe asthma exacerbations (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | during 52 weeks prior to inclusion
  Severe asthma exacerbation is defined as worsening of asthma requiring any of the following:
  * use of systemic corticosteroids (CS) (or a temporary increase in a stable OCS background dose) for at least 3 days or a single depo-injectable dose of CS and/or
  * an emergency room/urgent care visit (defined as evaluation and treatment for < 24 hours in an emergency department or urgent care center) due to asthma that required systemic CS (as per above) and/or
  * an inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥ 24 hours) due to asthma that required systemic CS.
7. Annualised rate of severe asthma exacerbations (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | during 52 weeks prior to inclusion
8. Cumulative days of severe asthma exacerbations (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | during 52 weeks prior to inclusion
9. Proportion of patients experiencing 0, 1, 2, ≥3 severe asthma exacerbations (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | 12 weeks
10. Proportion of patients with healthcare resource utilization (HRU) events (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | during 52 weeks prior to inclusion
  1. Unscheduled outpatient visits;
  2. Emergency department visits/emergency calls;
  3. Hospitalizations
11. Proportion of patients with HRU events (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | 12 weeks
  d. Unscheduled outpatient visits; e. Emergency department visits/emergency calls; f. Hospitalizations.
12.a Change from baseline in mean parameters of lung function at visit 2 (in case of availability of spirometry data) in all patients and in the cohort of patients receiving FDC budesonide/salbutamol | 12 weeks
  a. Pre- and post-FEV1 (Forced Expiratory Volume in 1 second). % predicted and L
12.b Change from baseline in mean parameters of lung function at visit 2 (in case of availability of spirometry data) in all patients and in the cohort of patients receiving FDC budesonide/salbutamol | 12 weeks
  b. Pre- and post-FVC (Forced Vital Capacity) (L)
12.c Change from baseline in mean parameters of lung function at visit 2 (in case of availability of spirometry data) in all patients and in the cohort of patients receiving FDC budesonide/salbutamol | 12 weeks
  c. Pre-FEF (Forced Expiratory Flow). Measured in L/sec.
Proportion of patients with controlled and partlly controlled asthma (in all patients and in the cohort of patients receiving FDC budesonide/salbutamol) | at inclusion into the study, then in 3 months (+-7days) after the inclusion
  according to the bronchial asthma symptom control questionnaire (ACQ-5). Uncontrolled asthma is defined as >1.5 points according to the Asthma Symptom Control Questionnaire (ACQ-5). The higher the score, the worse
To describe the Proportion of patients with history of smoking/current smokers at visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  applicable to smoking tobacco and electronic cigarettes (vapes)), and proportion of patients with change of smoking status at visit 3 compared to baseline (non-smoker/former smoker switched to current smoker, current smoker switched to former smoker);
To describe mean smoking index for current (tobacco) smokers, according to the assessment at visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  Mean smoking index to be evaluated in pack-years
To describe mean duration of smoking (years) for current e-cigarette (vape) smokers in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  according to the assessment at visit 3
To describe change of body mass index (BMI) to visit 3 compared to baseline in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  according to the assessment at visit 3
To describe proportion with overweight (BMI ≥25 kg/m2) in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe Change of body mass index (BMI) to visit 3 compared to baseline in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe proportion of patients with controlled and partly controlled asthma (according to GINA score) at visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe Proportion of patients with controlled and partly controlled asthma (according to the questionnaire ACQ-5) at visit 3 in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe Proportion of patients receiving FDC budesonide/salbutamol as monotherapy or in combination with basic therapy in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe Asthma therapy regimen from which the patient was switched to the FDC budesonide/salbutamol in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at visit 3;
To describe Proportion of patients with changes of inhaled asthma therapy occurred from visit 2 to visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  1. Change of basic therapy drug;
  2. Change of dose of basic therapy drug;
  3. Change of number of basic therapy drug inhalations per day;
  4. Change of ICS;
  5. Dose of ICS increased;
  6. Changes of another drug for maintenance therapy;
  7. Change in the type of drug delivery within the same INN (e.g. from capsule to powder or from aerosol to powder, etc.).
To describe Proportion of patients with OCS prescription occurred from visit 2 to visit 3; for patients already used OCS at visit 2 dose change will be evaluated in the cohort of patients receiving FDC budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe Proportion of patients with ICS-containing therapy as reliever and as maintenance at visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe number of budesonide/salbutamol inhalers used between visit 2 and visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe number of budesonide/salbutamol inhalations per month for a period from visit 2 to visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe proportion of patients experiencing 0, 1, 2, ≥3 severe asthma exacerbations* between visit 2 and visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe proportion of patients with HRU events occurred between visit 2 and visit 3 in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  1. Unscheduled outpatient visits;
  2. Emergency department visits/emergency calls;
  3. Hospitalizations.
To describe change from Visit 2 Pre- and post-FEV1 at visit 3 (in case of availability of spirometry data) in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe change from Visit 2 Pre- and post-FVC at visit 3 (in case of availability of spirometry data) in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3
To describe change from Visit Pre-FEF at visit 3 (in case of availability of spirometry data) in the cohort of patients receiving fixed-dose combination (FDC) budesonide/salbutamol on Visit 2 | 24 weeks
  assessment at Visit 3

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - Research Site, Gatchina
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Lipetsk
  - Research Site, Makhachkala
  - Research Site, Moscow
  - Research Site, Nizhny Tagil
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Tula
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org